CLINICAL TRIAL: NCT04884867
Title: "Sống Vui, Live Happily": A Psychosocial Tele-health Intervention to Address Multi-level Stigma Among Youth Living With HIV in Vietnam
Brief Title: A Psychosocial Tele-health Stigma Intervention for Youth Living With HIV in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Collaborators: Institute for Social Development Studies (ISDS) (Unknown); Fogarty International Center of the National Institute of Health (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mary DeSilva, Associate Research Professor, University of New England
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R21TW011085-01 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hiv; Stigma, Social
Keywords: HIV; Stigma; Vulnerable groups; Vietnam
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Social Stigma

STUDY DESIGN:
Masking Description: Participants will use a wireless pill container to monitor their adherence passively. Participants, lay coaches, and clinicians will all be blinded to adherence monitoring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive life skills coaching (Experimental): CBT-based supportive like skills delivered by phone by lay coaches
  Interventions: Behavioral: CBT-based supportive skills delivered by phone by lay coaches

INTERVENTIONS:
Behavioral: CBT-based supportive skills delivered by phone by lay coaches — 8-10 weekly coaching sessions delivered by telephone

SUMMARY:
The overall goals of the study are to deepen understanding of the spectrum of stigma experienced by YLHIV in Vietnam, to develop a multi-level stigma intervention for YLHIV delivered by telephone, and to evaluate the feasibility, acceptability, and preliminary efficacy of the intervention on intra- and inter-personal stigma, psychological wellbeing, and treatment adherence.

The project has the following Specific Aims:

1. Adapt a psychosocial stigma-reduction intervention for YLHIV in Vietnam based on cognitive-behavioral therapy principles and delivered by telephone, using input from youth during intervention development.
2. Assess the feasibility, acceptability and preliminary efficacy of this innovative approach to reduce stigma, and improve psychosocial wellbeing and ART adherence among YLHIV through a small pre-post study.
3. Explore the multiple facets of stigma experienced by YLHIV in Vietnam and their relationships with ART adherence and psychosocial wellbeing via quantitative surveys and electronic adherence monitoring.

The study will assess the feasibility and acceptability of this approach among YLVIV in Vietnam, and generate preliminary evidence for the potential effect of the intervention on important endpoints including stigma, psychosocial wellbeing, adherence, CD4 count, and viral load (VL).

DETAILED DESCRIPTION:
For the pilot, the investigators will recruit YLHIV on ART who self-report intrapersonal stigma and implement a 12-week pre-post intervention study in which participants will receive the phone-based intervention developed in the first phase. YLHIV will use an electronic adherence monitoring device for their ART medications.

In the pre-post intervention study, each of 40 patients will be followed for a total of 16 weeks. All patient subjects will be given an eCAP wireless pill container (WPC) that will be used to measure their adherence throughout the 16-week period. Study participation will involve two phases, with the following activities:

I. Adherence monitoring, pre-intervention period (Weeks 1-2). Once enrolled, the investigators will provide each subject with a WPC and instruction on correct use. The investigators will select one medication for each WPC. While subjects continue to receive care as usual, the investigators will collect their adherence data using the WPC.

II. Intervention period (Weeks 3-12). The intervention will be implemented for about 10 weeks; adherence data will be collected via WPCs through Week 16. They will remain blinded to the adherence information generated by the devices, as will their care providers.

ELIGIBILITY:
Inclusion Criteria:

* are between 18 and 24 years old
* are a patient at the OPC
* are expected to remain in care at the OPC for 3 months minimum(?)
* are currently on ART
* have primary responsibility for taking their own medications,
* self-report intrapersonal stigma via a brief screening questionnaire,
* are able to complete a short phone call from the location where they intend to be when participating in coaching sessions,
* agree to follow all study procedures, AND
* provide informed consent.

Exclusion Criteria:

* are below the age of 18 years or above the age of 24,
* are not currently on ART,
* live outside the clinic catchment area,
* are identified as having severe mental health issues as identified through screening, OR
* are not willing to provide informed consent.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Intrapersonal (self) Stigma | change between Week 1-Week 12
  modified 21-item self stigma subscale of Vietnam Stigma Index Studies instrument (People living with HIV: Stigma Index 2014; higher score=worse outcome)
Interpersonal Stigma | change between Week 1 and Week 12
  modified 21-item enacted stigma subscale of Vietnam Stigma Index Studies instrument (People living with HIV: Stigma Index 2014; higher score=worse outcome)
Depression | change between Week 1 and Week 12
  7-item depression subscale of the Depression, Anxiety and Stress Scale (DASS-21; higher score=worse outcome)
Anxiety | change between Week 1 and Week 12
  7-item depression subscale of the Depression, Anxiety and Stress Scale (DASS-21; higher score=worse outcome)
Adherence | Week 12 (endline)
  %≥95% on-time adherence

CONTACTS AND LOCATIONS:
Overall Officials: Mary DeSilva, ScD, MS, Principal Investigator — University of New England
Locations (1):
- Institute for Social Development Studies, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided